CLINICAL TRIAL: NCT01293344
Title: Gender Differences in Response to the Mediterranean Diet
Brief Title: Effects of the Mediterranean Diet on Cardiovascular Risk Profile in Men and Women
Acronym: ALIMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Simone Lemieux, Professor, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALIMED-2007-180 A3 R-2
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases; Controlled nutritional intervention; Sex differences; Women; Men; Cardiovascular risk; Lipid profile; Blood pressure; Insulin sensitivity; Inflammatory markers; Endothelial function; Oxidative stress
MeSH Terms: conditions — Cardiovascular Diseases; Multiple Endocrine Neoplasia Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Men and Mediterranean diet (Experimental): Men who are assigned to a 4 weeks experimental diet formulated to be concordant with characteristics of the traditional Mediterranean diet.
  Interventions: Other: Controlled nutritional intervention based on the Mediterranean diet
- Women and Mediterranean diet (Experimental): Women who are assigned to a 4 weeks experimental diet formulated to be concordant with characteristics of the traditional Mediterranean diet.
  Interventions: Other: Controlled nutritional intervention based on the Mediterranean diet

INTERVENTIONS:
Other: Controlled nutritional intervention based on the Mediterranean diet — Men are assigned to a 4 weeks isocaloric controlled nutritional intervention based on the Mediterranean diet (MedDiet) in which all foods and drinks are provided. The respective percentages of kcal derived from lipids, carbohydrates, protein and alcohol are respectively of 32%, 48%, 15% and 5%. Habitual energy intake of each participant is established by averaging energy requirements estimated by a validated food-frequency questionnaire (FFQ) and energy needs as determined by the Harris-Benedict formula. Body weight is measured on weekdays and total energy provided is revised if necessary for minimizing body weight fluctuations. This intervention period is preceded by a 4 weeks uncontrolled run-in period based on the Canada's Food Guide.
  Arms: Men and Mediterranean diet
Other: Controlled nutritional intervention based on the Mediterranean diet — Women are assigned to the same intervention than men in order to compare men and women metabolic response to the MedDiet.
  Arms: Women and Mediterranean diet

SUMMARY:
The purpose of this study is to document differences between men and women in changes in metabolic variables associated with cardiovascular risk in response to a 4 weeks isocaloric controlled nutritional intervention based on the Mediterranean diet in which all foods and drinks are provided to subjects. The investigators hypothesize that the decrease in LDL-cholesterol will be more important in men than in women.

DETAILED DESCRIPTION:
Nutritional interventions promoting the adoption of the traditional Mediterranean diet (MedDiet) are known to have significant and beneficial effects on cardiovascular disease (CVD) risk profile. On the other hand, recent evidence suggests that women respond differently to diet than men. No study has yet compared men and women metabolic response to the MedDiet in a controlled metabolic context in which all foods and drinks consumed are provided to the participant prepared by the research team. Therefore, we do not know whether being fed a MedDiet in controlled conditions would have similar health benefits in men and women. The purpose of this study is to document differences between men and women in changes in metabolic variables associated with cardiovascular risk in response to a 4 weeks isocaloric controlled nutritional intervention based on the MedDiet in which all foods and drinks are provided to subjects. We hypothesize that the decrease in LDL-cholesterol will be more important in men than in women. In this parallel controlled trial, both men and women are assigned to the same 4 weeks experimental diet formulated to be concordant with characteristics of the traditional MedDiet. Data will be collected before and after the controlled nutritional intervention based on the MedDiet.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopausal women from de Quebec City metropolitan area.
* Slightly elevated LDL-cholesterol concentrations (3.4-4.9 mM) or total cholesterol to HDL-C ratio ≥ 5.0
* At least one of the four following factors of the metabolic syndrome: 1) waist circumference > 94 cm in men and > 80 cm in women; 2) TG > 1.7 mmol/L; 3) fasting glycemia between 6.1 and 6.9 mmol/L and 4) blood pressure concentrations ≥ 130 / 85 mm Hg.
* Age: between 25 to 50 years
* Stable body weight (+/- 2.5 kg) for at least 3 months before the beginning of the study
* In women, a regular menstrual cycle for the last 3 months

Exclusion Criteria:

* Subjects with endocrine disorders, cardiovascular events, type 1 or 2 diabetes and those using medication that could affect dependent variables measured (namely lipid-lowering, hypoglycemic, insulin sensitizers and anti hypertensive medication)
* Smokers
* Subjects with history of alcoholism
* Subjects with food allergies or food aversion that could impede compliance to the Mediterranean diet
* Pregnant women and those using systemic hormonal contraceptives

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic outcomes | At baseline (at the beginning of the intervention) and at the end of the intervention period (4 weeks).
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, apolipoprotein (apo) B, apo A-1 and apo A-2 plasma concentrations, systolic and diastolic blood pressure, glucose and insulin concentrations during a 180-min oral glucose tolerance test, insulin sensitivity, CRP and Interleukine-6 levels, oxidized-LDL, E-selectin, ICAM-1 and VCAM-1.

SECONDARY OUTCOMES:
Nutritional variables | At baseline (at the beginning of the intervention), at the end of the intervention period (4 weeks) and at 6-months post-intervention (28 weeks).
  Dietary intakes
Eating behaviors | At baseline (at the beginning of the intervention) and at the end of the intervention period (4 weeks)
  Restraint, disinhibition, and susceptibility to hunger
Appetite ratings | At baseline (at the beginning of the intervention) and at the end of the intervention period (4 weeks)
  Desire to eat, hunger, fullness, and prospective food consumption
physical activity habits | At baseline (at the beginning of the intervention) and at the end of the intervention period (4 weeks)
  Weekly questionnaire about physical activities, a validated 3-day physical activity record (two weekdays and one weekend day)
Anthropometric measurements | At baseline (at the beginning of the intervention), at the end of the intervention period (4 weeks) and at 6-months post-intervention (28 weeks)
  Height, weight, body mass index, waist and hip circumferences,

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lemieux, Ph.D., Dt.P., Principal Investigator — Department of food sciences and nutrition / Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceuticals and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bedard A, Lamarche B, Corneau L, Dodin S, Lemieux S. Sex differences in the impact of the Mediterranean diet on systemic inflammation. Nutr J. 2015 May 12;14:46. doi: 10.1186/s12937-015-0035-y. PMID 25962728
- [Derived] Bedard A, Corneau L, Lamarche B, Dodin S, Lemieux S. Sex-related differences in the effects of the mediterranean diet on glucose and insulin homeostasis. J Nutr Metab. 2014;2014:424130. doi: 10.1155/2014/424130. Epub 2014 Oct 9. PMID 25371817
- [Derived] Bedard A, Tchernof A, Lamarche B, Corneau L, Dodin S, Lemieux S. Effects of the traditional Mediterranean diet on adiponectin and leptin concentrations in men and premenopausal women: do sex differences exist? Eur J Clin Nutr. 2014 May;68(5):561-6. doi: 10.1038/ejcn.2014.27. Epub 2014 Mar 5. PMID 24595221
- [Derived] Bedard A, Dodin S, Corneau L, Lemieux S. Impact of the traditional Mediterranean diet on the Framingham risk score and the metabolic syndrome according to sex. Metab Syndr Relat Disord. 2014 Mar;12(2):95-101. doi: 10.1089/met.2012.0076. Epub 2014 Jan 17. PMID 24438432